CLINICAL TRIAL: NCT04922710
Title: Physical Exercise for Augmenting Cognitive Health
Brief Title: Physical Exercise for Augmenting Cognitive Health (PEACH)
Acronym: PEACH
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study protocol was not feasible. We made several modifications but halted the study prematurely before we met our target sample size goal.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kirk Erickson, PhD, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20120192; R24AG065174-01 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Aging; Adverse Childhood Experiences
Keywords: Adverse Childhood Experiences; Brain Health; Cognitive Aging; Exercise; Reversibility Network
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A single group assigned a remote exercise intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based aerobic exercise (Experimental): Un-supervised exercise will be held 3 times a week for 60 minutes in the participant's home. Those who are unable to do a 60-minute session would instead complete it in two 30-minute sessions to reach the goal of exercising 150 minutes per week.
  Interventions: Behavioral: Home-based aerobic exercise

INTERVENTIONS:
Behavioral: Home-based aerobic exercise — Guidelines for exercise programming (ACSM, 2018) will be followed including a warmup and cool down, progressive and gradual increments in duration, and instruction regarding avoidance of physical activity related injury. The exercise group will receive moderate to vigorous intensity aerobic exercise for 60 minutes per day, three times a week, for 12 weeks. Participants who are unable to do a 60-minute session would instead complete it in two 30-minute sessions. The prescribed intensity will be based on estimated heart rate reserve, calculated using resting heart rate and age-adjusted heart rate maximum (220-age in years). Participants will maintain a minimum heart rate from their specific calculation that will be monitored by Polar Heart Rate straps.

SUMMARY:
PEACH is a pilot project which is being conducted to determine the feasibility and acceptability of a 12-week home-based exercise intervention among Black and African American adults. A secondary aim of the project is to determine whether the exercise intervention improves cognitive and psychological functioning.

DETAILED DESCRIPTION:
This pilot project aims to address the impact of early life adversity (ELA) on brain health in adulthood by conducting a pilot 12-week physical activity (PA) intervention delivered remotely using aerobic exercise bikes programmed to connect users with a trainer via an app. Investigators will recruit Black and African American individuals between the ages of 30-55 years (N = 40) who are currently sedentary and report experiencing at least one form of ELA prior to the age of 10. This study will be conducted at two sites: the University of Pittsburgh in Pittsburgh, PA, USA and the University of the West Indies in Kingston, Jamaica (site investigator: Terrence Forrester). At baseline and following the 12-week intervention, Investigators will collect a harmonized battery of cognitive, behavioral and psychosocial measures. The intervention itself will be home-based and will involve three 60-minute sessions of aerobic exercise per week using a Bluetooth-enable exercise bike. Participants' exercise programs will be supervised remotely by an exercise trainer and individualized depending on their age-adjusted heart rate reserve, with the goal being to have participants reach 50 minutes of moderate to vigorous intensity exercise per session by the end of the first 4 weeks of the intervention. The bikes will be outfitted with a tablet featuring an application called Neotiv. The Neotiv application will collect data from the bike regarding timing, duration, and intensity of exercise sessions, which will be securely shared with the exercise trainer to monitor attendance and adherence. The primary goals of this study are to determine whether the home-based exercise program (1) is feasible and acceptable (as measured by adherence and attendance), and (2) promotes improvements in cognitive and psychological functioning among adults who have been exposed to ELA, contingent on the feasibility. We realized that placing the health-related outcomes as primary or secondary outcomes would only make sense if the approach was feasible. Therefore, we revised the primary and secondary outcome measures to reflect the feasibility of the home-based exercise intervention program in terms of adherence and attendance.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 30-55 years
2. exposure to at least one form of threat-related adversity (e.g., exposure to violence; physical abuse) occurring prior to age 10 as documented by retrospective self-report
3. Self-identified Black or African American Race
4. access to high-speed internet
5. sedentary lifestyle (<60 minutes of PA/week).
6. no difficulties with mobility
7. Does not currently require the use of an assisted walking device
8. Does not have a history of balance difficulties
9. Not currently pregnant or planning to become pregnant in the next 12 months

Exclusion Criteria:

1. Psychosis
2. Significant suicide risk (i.e., current, active suicidal ideation with a plan)
3. Engaging in moderate-intensity exercise >=20 min per day, >=3 times per week
4. Current treatment for cancer
5. Neurological condition (MS, Parkinson's, Dementia, MCI) or brain injury (Stroke)
6. Substance use disorder in the past 3-months
7. Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep vein thrombosis (DVT) or other cardiovascular event
8. Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year
9. Sensory Impairment that would preclude neuropsychological testing
10. Not fluent in English
11. Travelling consecutively for 2+ weeks during the study
12. uncontrolled hypertension
13. Insulin-Dependent Diabetes Mellitus
14. Self-identified race anything other than Black or African American
15. Currently pregnant or planning to become pregnant in the next 12 months

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk I Erickson, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- Sennott Square, Pittsburgh, Pennsylvania, United States
- University of the West Indies, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
The data from this study will be made available to outside investigators under a data-sharing agreement. The data will be available to outside investigators after publication of the primary aims and at completion of quality control assessments and data organization. The investigators expect that the data from this study will result in interest from internal and external investigators for secondary analysis and ancillary projects.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Will be made available after study investigators have published summary data and primary aims results. Will be available for unlimited amount of time.
Access Criteria: Data requests will be approved by the PI and Co-PIs.

RESULTS

PARTICIPANT FLOW:
Groups:
- Home-based Aerobic Exercise: Un-supervised exercise will be held 3 times a week for 60 minutes in the participant's home
  Home-based aerobic exercise: Guidelines for exercise programming (ACSM, 2018) will be followed including a warmup and cool down, progressive and gradual increments in duration, and instruction regarding avoidance of physical activity related injury. The exercise group will receive moderate to vigorous intensity aerobic exercise for 60 minutes per day, three times a week, for 12 weeks. The prescribed intensity will be based on estimated heart rate reserve, calculated using resting heart rate and age-adjusted heart rate maximum (220-age in years). Participants will maintain a minimum heart rate from their specific calculation that will be monitored by Polar Heart Rate straps.
Period: Overall Study
Arm/Group | Home-based Aerobic Exercise
Started | 5 (Based on our IRB, 'enrolled' is anyone who signed the consent form even if they were screened ineligible after signing the consent form. So, 8 study participants signed the consent form and were 'enrolled'. Of these 8 subjects, 5 completed all the baseline outcome measures, met eligibility criteria and were subsequently assigned to receive the intervention.)
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Home-based Aerobic Exercise
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.40 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Exercise Intervention Program: Average Minutes Spent in Moderate to Vigorous Exercise
Description: Data regarding the average number of minutes spent engaging in moderate to vigorous exercise (via heart rate monitoring and comparison of heart rate to calculations based on heart rate reserve) will be collected to operationalize adherence. Adherence will be used as a metric of feasibility and acceptability.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Home-based Aerobic Exercise: Un-supervised exercise will be held 3 times a week for 60 minutes in the participant's home. Those who are unable to do a 60-minute session would instead complete it in two 30-minute sessions to reach the goal of exercising 150 minutes per week.
  Home-based aerobic exercise: Guidelines for exercise programming (ACSM, 2018) will be followed including a warmup and cool down, progressive and gradual increments in duration, and instruction regarding avoidance of physical activity related injury. The exercise group will receive moderate to vigorous intensity aerobic exercise for 60 minutes per day, three times a week, for 12 weeks. The prescribed intensity will be based on estimated heart rate reserve, calculated using resting heart rate and age-adjusted heart rate maximum (220-age in years). Participants will maintain a minimum heart rate from their specific calculation that will be monitored by Polar Heart Rate straps.
Arm/Group | Home-based Aerobic Exercise
Number analyzed (Participants) | 4
Minutes | 1578.5 (721.73)

2. Secondary Outcome: Adherence to Exercise Intervention Program: Number of Sessions Completed
Description: Data regarding the number of exercise sessions completed will be collected to operationalize adherence. Adherence will be used as a metric of feasibility and acceptability.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Number of sessions
Arm/Group | Home-based Aerobic Exercise
Number analyzed (Participants) | 4
Number of sessions | 51.25 (13.15)

3. Other Pre Specified Outcome: Mean Change in Systolic Blood Pressure
Description: Systolic blood pressure (SBP) will be measured at baseline and 12-weeks to determine whether there is a change in SBP.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Mean Change in Physical Activity
Description: Participants will complete one week of actigraphy at baseline and again at follow-up to determine whether physical activity levels change. This will be operationalized as change in average number of steps per day.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Mean Change in Heart Rate
Description: Heart rate will be measured throughout the intervention and changes in heart rate from baseline to the end of the intervention will be calculated.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percent Change in Total Body Weight
Description: Participants will be weighed on a calibrated stadiometer both before and after the intervention. The investigators will examine percent changes in body weight before and after the intervention.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mean Change in Negative and Positive Affect
Description: This will be calculated via scores from the Positive and Negative Affect Scale. Scores can range from 1 to 100, with 1 meaning less positive affect and 100 meaning more positive affect.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Mean Change in Depressive Symptoms
Description: Participants will complete the Center for Epidemiological Studies-Depression Scale, a measure of the frequency of 20 common depressive symptoms rated along a 0 ("rarely or none of the time") to 3 ("most or all of the time") Likert scale. Responses are summed to yield a total symptom score (maximum possible score of 60) with higher scores reflecting more severe depressive symptoms.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Change in Perceived Stress
Description: Participants will complete the Perceived Stress Scale (PSS) a measure of the frequency of 20 common depressive symptoms rated along a 0 ("rarely or non, a 14-item measure that assesses experiences of daily life stress. The PSS is an instrument on which respondents use a 0 ("never") to 4 ("very often") Likert scale to rate the degree to which daily life events are perceived to be uncontrollable, unpredictable, or unmanageable. Responses are summed to form a total score (maximum possible score of 56).
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Change in Picture Sequence Performance
Description: A Picture Sequence task will be administered at baseline, and then following the intervention (12-weeks). The main outcome from this task is the cumulative number of adjacent pictures in which a participant correctly remembered the sequence. A lower number of correct items indicates worse episodic memory.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Mean Change in Picture Vocabulary Performance
Description: A Picture Vocabulary task will be administered at baseline, and then following the intervention (12-weeks). Participants will be presented with visual stimuli along with an auditory cue and will have to judge which of the visual stimuli match the auditory cue. The main outcome from this task is total items answered correctly, with a lower number of items being indicative or worse language ability.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mean Change in Pattern Comparison Performance
Description: A Pattern Comparison task will be administered at baseline, and then following the intervention (12-weeks). Participants will be presented with visual patterns and asked to respond whether the patterns are the same or different. The main outcome from this task is total items answered correctly in the 90 seconds allotted for the task, with a lower number of items being indicative or worse processing speed.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Adherence to Exercise Intervention Program: Average Duration of Sessions
Description: Data regarding the average duration of sessions will be collected to operationalize adherence. Adherence will be used as a metric of feasibility and acceptability.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Change in Flanker Performance
Description: A Flanker task will be administered at baseline, and then following the intervention (12-weeks). The main outcome from this task is an interference effect (in ms) which indicates how much longer it takes for a participant to make a directional response to a center arrow when the flanking arrows are arranged in congruent vs. incongruent direction from the center stimulus. A higher interference effect indicates worse executive functioning.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Mean Change in Dimensional Card Sort Performance
Description: A Dimensional Card Sort task will be administered at baseline, and then following the intervention (12-weeks). The main outcome from this task is an interference effect (in ms) which indicates how much longer it takes for a participant to match a stimulus to other choice stimuli based on a feature (shape or color), with the feature participants must match on switching without warning during the task. A higher interference effect indicates worse executive functioning.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mean Change in List Sorting Performance
Description: A List Sorting task will be administered at baseline, and then following the intervention (12-weeks). Participants will be presented with a series of stimuli and then be asked to repeat the stimuli in order of size from smallest to largest. The main outcome from this task is total items answered correctly, with a lower scoring being indicative or worse working memory.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: In this exercise intervention, there is no expected long-term risk for serious adverses or all-cause mortality.
Arm/Group | Home-based Aerobic Exercise
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04922710/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04922710/ICF_001.pdf